CLINICAL TRIAL: NCT01493180
Title: Exploratory Study of OPC-12759 Ophthalmic Suspension in Patients With Keratoconjunctiva Epithelial Disorder
Brief Title: Exploratory Study of OPC-12759 Ophthalmic Suspension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 037E-11-002; JapicCTI-111708 (Other: Japic)
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Results first posted 2014-03-03 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-02

CONDITIONS: Keratoconjunctival Epithelial Disorder

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OPC-12759 ophthalmic suspension (Experimental): OPC-12759 ophthalmic suspension
  Interventions: Drug: OPC-12759 ophthalmic suspension
- Sodium hyaluronate ophthalmic solution (Active Comparator): Sodium hyaluronate ophthalmic solution
  Interventions: Drug: Sodium hyaluronate ophthalmic solution

INTERVENTIONS:
Drug: OPC-12759 ophthalmic suspension — OPC-12759 ophthalmic suspension 2%
  Arms: OPC-12759 ophthalmic suspension
Drug: Sodium hyaluronate ophthalmic solution — Sodium hyaluronate ophthalmic solution 0.1%
  Arms: Sodium hyaluronate ophthalmic solution

SUMMARY:
The purpose of this study is to evaluate the efficacy of OPC-12759 ophthalmic suspension for patients with keratoconjunctival epithelial disorder compared with sodium hyaluronate. Also, safety of OPC-12759 is to be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of superficial punctate keratopathy, corneal erosion or persistent epithelial defect
2. Fluorescein corneal staining score of 3 or higher

Exclusion Criteria:

1. Active ocular infection
2. Vernal keratoconjunctivitis
3. Recurrent corneal erosion
4. Physical irritation of eyelashes or relaxed bulbar conjunctiva to cornea or conjunctiva
5. Subjects who cannot discontinue or anticipate use of eye drops except for limited concomitant ones during the study. Soft-santear is allowed during the screening period.
6. Anticipated use of contact lens during the study.
7. Insertion of punctal plug or fall out of punctal plug within 3 months
8. Subjects who are judged by the investigator to be ineligible for the study because of a past or concurrent systemic disease.
9. Receipt of any investigational product within 4 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-12; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eiji Murakami, Study Director — Division Dermatilogicals and Ophtalmolgicals, Otsuka Pharmaceutical Co., Ltd.
Locations (10):
- Japan (10):
  - Kanto region, Hachiōji
  - Kansai region, Ibaraki
  - Kansai region, Ikoma
  - Kansai Region, Kobe
  - Chugoku region, Kure
  - Kansai region, Kyoto
  - Tokai region, Nagoya
  - Kansai region, Osaka
  - Kansai region, Sayama
  - Kanto region, Tokyo

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OPC-12759 Ophthalmic Suspension | Sodium Hyaluronate Ophthalmic Solution
Started | 51 | 51
Completed | 48 | 49
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OPC-12759 Ophthalmic Suspension | Sodium Hyaluronate Ophthalmic Solution | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (17.9) | 54.5 (20.9) | 54.7 (19.3)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 27 | 58
  >=65 years | 20 | 24 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 34 | 75
  Male | 10 | 17 | 27
Region of Enrollment [Number; unit: participants]
  Japan | 51 | 51 | 102

OUTCOME MEASURES:

1. Primary Outcome: Change in the Keratoconjunctival Staining Score From Baseline
Description: Keratoconjunctival staining indicates the damage to the corneal and conjunctival epithelium. The cornea and conjunctiva were divided into 3 and 2 fractions, respectively, each of which was given a staining score from 0 to 3, and the total score was calculated (0-15). 0 is better.
  The change from baseline at the end of instillation (LOCF) in the keratoconjunctival staining score were compared between the 2% rebamipide group and the 0.1% sodium hyaluronate group using a t-test.
Time Frame: Basekine, 4 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | OPC-12759 Ophthalmic Suspension | Sodium Hyaluronate Ophthalmic Solution
Number analyzed (Participants) | 51 | 51
scores on a scale | -3.4 (2.7) | -3.1 (2.4)
Statistical Analysis 1: Comparison: OPC-12759 Ophthalmic Suspension vs Sodium Hyaluronate Ophthalmic Solution; Test type: Superiority or Other; p = 0.576, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | OPC-12759 Ophthalmic Suspension | Sodium Hyaluronate Ophthalmic Solution
Serious Adverse Events (participants affected / at risk) | 1/51 | 0/51
Other Adverse Events (participants affected / at risk) | 16/51 | 12/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OPC-12759 Ophthalmic Suspension (N=51) | Sodium Hyaluronate Ophthalmic Solution (N=51)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OPC-12759 Ophthalmic Suspension (N=51) | Sodium Hyaluronate Ophthalmic Solution (N=51)
Chalazion (Eye disorders) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 3 (3) | 3 (3)
Corneal deposits (Eye disorders) | 1 (1) | 0 (0)
Corneal infiltrates (Eye disorders) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Punctate keratitis (Eye disorders) | 1 (1) | 0 (0)
Trichiasis (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysgeusia (bitter taste) (Nervous system disorders) | 4 (4) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vocal cord inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No